CLINICAL TRIAL: NCT03659019
Title: Follow-up Database of Patients Who Are Candidates for Implanted Phrenic Nerve Stimulator and Implanted Patients
Brief Title: Implanted Phrenic Nerve Stimulator Database.
Acronym: SPi-REG
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Neuroresp, Reference centre Syndrome d'Ondine (Unknown)
Responsible Party: Sponsor
Other Study IDs: NI17032J.
Record Dates: First submitted 2018-08-27; First posted 2018-09-06 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: External Mechanical Ventilatory Support

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ventilatory paralysis: dependence on mechanical ventilatory support
  Interventions: Other: Quality of life questionnaires
- central hypoventilation: documented permanent or nocturnal hypoventilation
  Interventions: Other: Quality of life questionnaires

INTERVENTIONS:
Other: Quality of life questionnaires — During 10 years, the study will be conduct to obtain the quality of life evolution and medical complications in patients candidates but not implanted, and in patients candidates then implanted with the phrenic nerve stimulator.

SUMMARY:
Phrenic nerve stimulation is a neurostimulation technique that allows patients who are dependent on external mechanical ventilatory support to regain their breathing autonomy. This study aim at long term following of patients who may be candidates for permanent implanted phrenic nerve stimulator.

DETAILED DESCRIPTION:
During 10 years, the study will be conduct to obtain the quality of life evolution and medical complications in patients candidates but not implanted, and in patients candidates then implanted with the phrenic nerve stimulator.

ELIGIBILITY:
Inclusion Criteria:

* Patients with central respiratory paralysis (medullary lesions or supramedullary lesions, whatever their causes) or patients with congenital central hypoventilation (including Ondine syndrome by Phox2B mutation) or acquired (whatever the cause), with permanent hypoventilation or related to sleep.

Exclusion Criteria:

* Patient not affiliated to the social security system
* Patient unable to oppose his participation in research
* Patient not understanding French

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients adressed to the Respiratory and Medical Resuscitation Unit of the Pitié-Salpêtrière Charles Foix Hospital Group for the search for an indication of SPi in the context of central ventilatory paralysis or central hypoventilation, whether or not the indication is retained at the end of the balance sheet; this population is essentially made up of adults, some but not all of whom benefit from a protection regime; it may occasionally include minors;
  Patients addressed to the adult branch of the Rare Disease Reference Center for Congenital Central Venous Hypoventilation, located within the hospital group Pitié-Salpêtrière Charles Foix, for the assessment and monitoring of their disease. By definition, this population consists solely of adults.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-11-20 (Actual); Primary Completion 2028-11-19 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Score at the Medical Outcomes Study Short-Form General Health Survey (SF-12) scale in patients with implanted phrenic nerve stimulator | 10 years
  Evolution of the physical (score between 9.95 and 70.02) and mental (score between 5.89 and 71.97) dimensions included into the SF-12 scale in patients with implanted phrenic nerve stimulator before, and up to 10 years after the implantation

SECONDARY OUTCOMES:
Number of evolving episodes involving care, whether pathology events or intercurrent events | 10 years
  Follow-up of complications in implanted patients compared with the natural course of the disease (i.e. non-implanted patients)

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas SIMILOWSKI, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No